CLINICAL TRIAL: NCT07353645
Title: Phase I/II Clinical Study of KRAS Neoantigen Nanovaccine as Adjuvant Therapy for Colorectal Cancer/Pancreatic Cancer With High Risk of Recurrence
Brief Title: KRAS Neoantigen Nanovaccine as Adjuvant Therapy for Colorectal Cancer/Pancreatic Cancer
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2025-1111-02
Record Dates: First submitted 2025-12-29; First posted 2026-01-20 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2025-12

CONDITIONS: Colorectal Cancer; Pancreatic Cancer
MeSH Terms: conditions — Colorectal Neoplasms; Pancreatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental Group (Experimental): neoantigen nanovaccine constructed from the bacterial membranes of engineered Lactococcus lactis, independently developed by the Cancer Center of Nanjing Drum Tower Hospital. It is administered via subcutaneous or intralymph node injection.
  Interventions: Drug: KRAS Neoantigen Nanovaccine

INTERVENTIONS:
Drug: KRAS Neoantigen Nanovaccine — The vaccine utilizes a neoantigen nanovaccine constructed from the bacterial membranes of engineered Lactococcus lactis, independently developed by the Cancer Center of Nanjing Drum Tower Hospital. It is administered via subcutaneous or intralymph node injection.
  Other Names: a PD-1/CTLA-4 bispecific antibody

SUMMARY:
This clinical trial will utilize a neoantigen nanovaccine constructed from the bacterial membranes of an engineered Lactococcus lactis strain (FOLactis). This platform, independently developed by our center, expresses KRAS antigenic peptides. The vaccine will be administered as adjuvant therapy to post-operative patients with colorectal or pancreatic cancer who carry KRAS mutations and are at high risk of recurrence. The study aims to assess the safety, immunogenicity, and preliminary efficacy of this neoantigen nanovaccine in a clinical setting.

DETAILED DESCRIPTION:
1. Pre-vaccination Screening: Detection of KRAS hotspot mutations in the patient's tumor tissue.
2. Vaccine Composition and Administration: The vaccine utilizes a neoantigen nanovaccine constructed from the bacterial membranes of engineered Lactococcus lactis, independently developed by the Cancer Center of Nanjing Drum Tower Hospital. It is administered via subcutaneous or intralymph node injection.

   The study consists of two phases: Dose Escalation and Dose Expansion. The Dose Escalation phase involves the vaccine alone, while the Dose Expansion phase combines the vaccine with a PD-1/CTLA-4 bispecific antibody, as detailed below:

   Dose Escalation Phase: Conducted according to a "3+3" design. The neoantigen nanovaccine is tested at two dose levels: 1.5mg and 3.0mg. Each injection has a total volume of 1.0ml, administered subcutaneously in the subdeltoid region of both upper arms and the lateral thigh muscle group, or via ultrasound-guided injection into bilateral inguinal lymph nodes. Vaccination Schedule: A total of 9 vaccinations are planned on Days 1, 4, 8, 15, 22, 43, 64, 85, and 106. Vaccinations #1 and #5-#9: Ultrasound-guided bilateral inguinal lymph node injection combined with subcutaneous injection in the subdeltoid region. Vaccinations #2, #3, and #4: Subcutaneous injection in the subdeltoid region and lateral thigh muscle group, accompanied by intravenous cyclophosphamide (200mg/m²) on the same day. Efficacy and Safety Monitoring: Radiographic efficacy evaluations are performed every 12 weeks for the first two years post-surgery, and every 24 weeks thereafter. Adverse events are assessed following each vaccination.

   Dose Expansion Phase: The vaccine dose for this phase is determined based on results from the Dose Escalation phase. The vaccination procedure remains the same. Twenty eligible post-operative colorectal cancer patients and twenty eligible post-operative pancreatic cancer patients will be enrolled for continued observation of efficacy and side effects. The nanovaccination schedule follows the Dose Escalation phase protocol. The PD-1/CTLA-4 bispecific antibody is administered starting on the first day of vaccination, once every three weeks, until disease progression, unacceptable toxicity, or completion of 18 cycles (approximately 1 year of treatment), whichever occurs first.
3. Immunological Follow-up: Hematological immune monitoring, including lymphocyte immunophenotyping and cytokine profiling, is performed pre-vaccination and on Days 1, 22, 43, 85, and 106 after the first vaccination.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years and ≤75 years, with an ECOG performance status of 0-1.
* Patients with histologically confirmed colorectal adenocarcinoma or pancreatic adenocarcinoma who have undergone radical resection (R0) and completed at least 4 cycles of postoperative adjuvant chemotherapy.
* Postoperative pathological stage for colorectal cancer is IIIA, IIIB, or IIIC. For pancreatic cancer, postoperative pathological stage is I, II, or III. The tumor must harbor at least one of the following KRAS hotspot mutations: G12D, G12V, G12R, G12A, G12S, G12C, or G13D.
* No radiological evidence of tumor recurrence or metastasis.
* Patients must meet the following hematologic criteria: Lymphocyte count ≥0.5×10⁹/L, neutrophil count ≥1.5×10⁹/L, white blood cell count >2.5×10⁹/L; Hemoglobin ≥90 g/L; Platelet count ≥90×10⁹/L.
* Patients must meet the following biochemical criteria: Total bilirubin ≤1.5 × upper limit of normal (ULN); AST and ALT ≤1.5 × ULN; Serum creatinine ≤1.5 × ULN or creatinine clearance ≥30 mL/min.
* Patients must meet the following coagulation criteria: INR or PTT ≤1.5 × ULN.
* Patients of childbearing potential must employ adequate contraception or other birth control methods before enrollment and throughout the trial.
* Signed informed consent form has been obtained.
* Ability to comply with the study protocol and follow-up procedures.

Exclusion Criteria:

* Patients with colorectal cancer exhibiting microsatellite instability-high (MSI-H)/deficient mismatch repair (dMMR) or harboring BRAF mutations.
* Pancreatic cancer patients with neuroendocrine tumor components are excluded.
* Patients with a history of other malignancies, except for carcinoma in situ of the cervix, treated squamous cell carcinoma or bladder epithelial tumors (Ta and TIS), or other malignancies that have been curatively treated (at least 5 years prior to enrollment).
* Prior treatment with anticancer vaccines or any antibodies targeting T-cell co-regulatory proteins (e.g., anti-PD1, anti-PDL1, or anti-CTLA4).
* Patients with HIV, HCV, or HBV infection; uncontrolled coronary artery disease or asthma; uncontrolled cerebrovascular disease; or any other condition deemed by the investigator as grounds for exclusion.
* Patients who are on immunosuppressants or systemic corticosteroid therapy for immunosuppressive purposes (at a dose >10 mg/day prednisone or equivalent) and have continued use within 2 weeks prior to enrollment.
* Poorly controlled cardiac clinical symptoms or diseases, such as: Heart failure of NYHA Class II or higher; Unstable angina; Myocardial infarction within the past year; Clinically significant supraventricular or ventricular arrhythmia requiring treatment or intervention; QTc >450 ms (males); QTc >470 ms (females).
* Abnormal coagulation function (INR >2.0, PT >16 s), bleeding tendency, or current thrombolytic or anticoagulant therapy. Prophylactic use of low-dose aspirin or low molecular weight heparin is allowed.
* Patients with active infection; unexplained fever ≥38.5°C within 7 days prior to medication; baseline white blood cell count >15×10⁹/L; or suppurative and chronic infections with non-healing wounds.
* Pregnant or lactating women. Women of childbearing potential must have a negative pregnancy test within 7 days prior to enrollment.
* Substance abuse, or clinical, psychological, or social factors that may affect the provision of informed consent or the conduct of the study.
* Known or suspected allergy to drugs used in immunotherapy.
* Inability to undergo immunological and clinical follow-up assessments.
* Known history of allogeneic organ transplantation or allogeneic hematopoietic stem cell transplantation.
* Participation in other interventional drug clinical trials concurrently.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Estimated)
Dates: Start 2026-01-10 (Estimated); Primary Completion 2029-01-01 (Estimated); Study Completion 2031-01-01 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicities (DLT) | From clinical trial enrollment until the date of first documented progression or date of death from any cause, whichever came first, assessed up to five years.

SECONDARY OUTCOMES:
Proportion of patients with a decrease in positive tumor markers (ctDNA and/or CEA/CA199) | 3 months post-first vaccination
Proportion of patients with clearance of positive tumor markers (ctDNA and/or CEA/CA199) | 3 months post-first vaccination
KRAS neoantigen specific T cells | From clinical trial enrollment until the date of first documented progression or date of death from any cause, whichever came first, assessed up to five years.
  From clinical trial enrollment until the date of first documented progression or date of death from any cause, whichever came first, assessed up to five years.
Recurrence-free survival (RFS) | From clinical trial enrollment until the date of first documented progression or date of death from any cause, whichever came first, assessed up to five years.
Correlation between neoantigen-specific T-cell frequency and dynamic changes in tumor markers (ctDNA and/or CEA/CA199) | From clinical trial enrollment until the date of first documented progression or date of death from any cause, whichever came first, assessed up to five years.
  Unit of Measure: Percent change in concentration (%) Measurement Tool/Description: The frequency of neoantigen-specific T cells (as a percentage of CD8+ T cells) quantified using multiparameter flow cytometry in peripheral blood or tumor microenvironment will be correlated (e.g., using Pearson or Spearman correlation coefficient) with the percent change in serum tumor marker levels (ctDNA and/or CEA/CA199).
Association between neoantigen-specific T-cell frequency and recurrence-free survival (RFS) | From the date of surgery/treatment initiation to the date of first documented disease recurrence or death from any cause. Assessment will be based on radiographic evaluation and clinical follow-up.
  Unit of Measure: Months Measurement Tool/Description: Assessment will be based on radiographic evaluation and clinical follow-up.The frequency of neoantigen-specific T cells (as a percentage of CD8+ T cells) quantified using multiparameter flow cytometry]in peripheral blood or tumor microenvironment will be correlated (e.g., using Pearson or Spearman correlation coefficient) with time in months from the date of surgery to the date of first documented disease recurrence or death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Baorui Liu, Study Chair — Nanjing Drum Tower Hospital Affiliated to Medical School of Nanjing University
Locations (1):
- Nanjing Drum Tower Hospital Affiliated to Medical School of Nanjing University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No